CLINICAL TRIAL: NCT07397429
Title: Group Therapy Using the I-Reconstruction Psychotherapy Method for Reducing Anxiety Levels: a Randomized Controlled Trial
Brief Title: Group Therapy Using the "I-Reconstruction" Psychotherapy Method to Reduce Anxiety Levels
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: International Association Psychosomatics And Health Therapy (Other)
Responsible Party: Principal Investigator, Tetiana Pavlenko, Research Director, author of the "I - reconstruction" method, Supervisor, International Association Psychosomatics And Health Therapy
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Onorul88
Record Dates: First submitted 2026-01-08; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Anxiety; Anxiety Depression
Keywords: Anxiety,; Group Therapy; Randomized Controlled Trial - RCT; Anxiety Disorders; Psychotherapeutic Intervention; Depression; I - Reconstruction; Internal Conflict Test; Preverbal trauma
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Standard of Care; Therapeutics

STUDY DESIGN:
Intervention Model Description: A Randomized Controlled Trial with three parallel groups (2 experimental and 1 control). The duration of participation is 12 months (10-session core course + follow-up assessments at 3, 6, and 12 months).
  This study will be conducted online, based at the International Association of Psychosomatics and Body Therapy. Participant recruitment will be conducted via social media and the Association's online platforms.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Given the nature of the intervention (an active, structured group psychotherapy "I-Reconstruction" compared to supportive group psychotherapy), full blinding of participants and therapists is not possible.
  However, to minimize the risk of bias and ensure methodological rigor, partial blinding will be applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active "I-Reconstruction" Therapy Group 1 (Experimental): Participants randomized to the experimental group received the active psychotherapeutic intervention "l-Reconstruction." This group consisted of adults with clinically significant anxiety who met all inclusion criteria of the study. Participants attended ten weekly online group therapy sessions led by a certified "l-Reconstruction" therapist. The group format was designed to facilitate therapeutic change through guided interpersonal interaction, normalization of experiences, and reflection within a structured therapeutic framework. All participants in the experimental group completed baseline, post-intervention, and follow-up assessments to evaluate changes in anxiety and related psychological outcomes.
  Interventions: Drug: Experimental: Active "I-Reconstruction" Therapy
- Active "I-Reconstruction" Therapy Group 2 (Experimental): Participants randomized to the experimental group received the active psychotherapeutic intervention "l-Reconstruction." This group consisted of adults with clinically significant anxiety who met all inclusion criteria of the study. Participants attended ten weekly online group therapy sessions led by a certified "l-Reconstruction" therapist. The group format was designed to facilitate therapeutic change through guided interpersonal interaction, normalization of experiences, and reflection within a structured therapeutic framework. All participants in the experimental group completed baseline, post-intervention, and follow-up assessments to evaluate changes in anxiety and related psychological outcomes.
  Interventions: Drug: Experimental: Active "I-Reconstruction" Therapy
- Control Group (Other): Standard Care (Treatment as Usual) Participants randomized to the control group received no therapeutic intervention during the study period. They continued with their usual daily activities and were not restricted from seeking any form of support or care outside the study. The control group participated only in scheduled psychological assessments at baseline, post-intervention, and follow-up time points, allowing for comparison of outcome trajectories between the intervention and non-intervention conditions.
  Interventions: Drug: Standard Care (Treatment as Usual)

INTERVENTIONS:
Drug: Experimental: Active "I-Reconstruction" Therapy — The intervention consisted of a structured group psychotherapy program based on the "l-Reconstruction" method. The program included ten weekly group sessions, each lasting 120 minutes, delivered online by a certified therapist trained in the method. The intervention targeted anxiety through therapeutic work with preverbal trauma and internal conflicts by reconstructing core personality components related to desire, ownership, and the capacity for pleasure. The therapeutic process combined psychoeducation, analysis of preverbal acts, exploration of emotional and bodily responses, reconstruction of traumatic experiential patterns, and structured group reflection and integration. The intervention followed a standardized protocol to ensure consistency across groups and therapists.
  Other Names: I-Reconstruction
  Arms: Active "I-Reconstruction" Therapy Group 1; Active "I-Reconstruction" Therapy Group 2
Drug: Standard Care (Treatment as Usual) — Participants assigned to the control group did not receive any structured psychotherapeutic intervention as part of the study. During the intervention period, no active treatment, group sessions, or therapeutic procedures were provided by the research team. The control condition was designed to serve as a non-intervention comparison group for evaluating the effects of the "l-Reconstruction" group psychotherapy.
  Arms: Control Group

SUMMARY:
Brief Summary of the Study The aim of this clinical trial is to find out if the group therapy method "Self-Reconstruction" helps to reduce anxiety in adults. The researchers want to see if the participants' emotional state becomes more stable after completing the course.

The main questions that this study aims to answer are:

Do people's anxiety levels decrease after taking the course of "I-Reconstruction" classes?

Do the positive effects of the classes persist 3, 6 and 12 months after they finish?

Do the participants' quality of life and ability to enjoy life improve?

The researchers will compare a group of people who attend the therapy classes with a group of people who receive usual care to see if the new method is more effective.

Participants will:

Participate in 10 online group meetings once a week.

Do simple breathing and movement exercises to calm the body and emotions.

Discuss your feelings and desires with a professional in a safe group.

Complete questionnaires about your condition at the beginning, during, and after the study.

DETAILED DESCRIPTION:
RESEARCH PROTOCOL (CONSORT) Title Group Therapy using the I-Reconstruction Psychotherapy Method for Anxiety Reduction: A Randomized Controlled Trial.

1. Rationale Anxiety disorders remain one of the most widespread forms of mental pathology, significantly reducing the quality of life and social functioning of millions of people worldwide. Despite the recognized efficacy of Cognitive Behavioral Therapy (CBT) and pharmacological treatment as empirically supported approaches, a significant percentage of patients do not achieve full remission, and the treatment gap remains critically large. This underscores the necessity for finding and empirically testing new, deep-rooted psychotherapeutic interventions. This is where the I-Reconstruction psychotherapy method becomes relevant.

   The I-Reconstruction method is a new but promising approach that offers a unique perspective on personality structure and the genesis of anxiety disorders. Central to the method are desire, possession, and satisfaction, which are viewed not merely as mental states but as fundamental structural elements of the personality that shape its interaction with the world. Dysfunctions or conflicts within these elements-specifically, impaired capacity to possess one's own emotional and life resources or the frustration of desire-directly lead to the formation of anxiety.

   From the perspective of modern psychology, the inability to achieve satisfaction or unfulfilled desire are often catalysts for anxiety and pathological fixation. Researchers emphasize that impairments in self-regulation processes, including the capacity for adequate desire and the attainment of satisfaction, are closely linked to the development of a wide range of mental disorders, including anxiety. Specifically, issues with self-esteem and the possession of internal states often manifest as generalized anxiety and avoidance, highlighting the need for psychotherapeutic intervention aimed at these deeper structures. While CBT focuses on cognitive and behavioral patterns, I-Reconstruction aims for deeper change by restoring the integration of desire and possession as a healthy foundation for obtaining satisfaction, which is theoretically expected to yield a more stable reduction in anxiety levels.

   Contemporary empirical studies confirm the link between this triad and the emergence of anxious symptoms. For instance, within Self-Determination Theory, the frustration of basic needs for autonomy and competence-i.e., the disruption of the sense of agency and possession over one's own actions-correlates with heightened anxiety and reduced psychological well-being. This mechanism demonstrates that the lack of experience in "possessing" one's own desires or internal states can intensify feelings of helplessness and loss of control-core characteristics of anxiety.

   Secondly, neuro- and psychophysiological studies indicate that reward system dysfunctions-reduced anticipation of reward and difficulties in experiencing pleasure (anhedonia)-are found not only in depression but are also associated with anxious manifestations. Research on reward processing shows that reduced reward sensitivity and changes in neural correlates of reward are linked to persistent tension, hypervigilance, and altered decision-making strategies that maintain anxious states.

   Thus, when desire remains frustrated, the sense of possession over one's experience is weakened, and the ability to experience satisfaction is impaired, a "triad of frustration" is formed that can sustain anxiety at cognitive, emotional, and bodily levels. This picture provides an empirical basis for applying the I-Reconstruction method, which aims to restore agency (possession), actualize conscious desires, and restore the capacity to experience satisfaction in order to stabilize anxious symptoms.
2. Design This study is a randomized controlled trial (RCT) with three parallel groups (2 experimental and 1 control). The duration of participation for each participant is approximately 17 months. This period includes a screening and initial assessment phase (T1), a course of therapy sessions (T2-T3), and a series of delayed measurements at 3, 6, and 12 months after the intervention (T4-T6).

2.1. Recruitment and selection process of participants Recruitment will be used online through the official pages of the NGO "International Association of Psychosomatics and Health Therapy" on social networks (Facebook, Instagram) and on the Association's website. An information announcement will be published with a description of the study, participation criteria and links to the screening survey.

Potential participants who express interest will be directed to an online questionnaire (implemented on the Google Forms platform), where they will fill in:

* Demographic data.
* Screening tools: Beck Anxiety Inventory (BAI), HADS-A anxiety subscale, Diagnosis of Preverbal Dysregulation (DPD) questionnaire and Internal Conflict Test (ICT) to check inclusion/exclusion crit

ELIGIBILITY:
Inclusion Criteria:

Age between 18 and 55 years (inclusive).

Clinically significant level of anxiety according to the Beck Anxiety Inventory (BAI) ≥ 9 points.

Anxiety subscale score on the Hospital Anxiety and Depression Scale (HADS-A) ≥ 11 points.

Significant level of preverbal trauma according to the "Diagnostics of Preverbal Dysregulation" (DPD, T. Pavlenko) questionnaire: total score ≥ 16.

Specific subscale scores in DPD: "Desire" ≥ 5, "Satisfaction" ≥ 5, and "Possession" (Obsession) ≥ 6 points.

Presence of internal conflicts according to the "Internal Conflict Test" (ICT) ≥ 1 point on the skin tissue measurement scale.

Willingness to comply with the study protocol and the online therapy format.

Exclusion Criteria:

Current participation in any other psychotherapy during the study.

Use of any psychotropic medications within the last 30 days (antidepressants, tranquilizers, neuroleptics, mood stabilizers).

Diagnosed severe mental disorders (according to ICD-10/DSM-5) requiring specialized psychiatric care or inpatient treatment.

Presence of acute suicidal risk.

Substance abuse (alcoholism, drug addiction).

Failure to meet any of the threshold values specified in the inclusion criteria.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-03-02 (Estimated); Primary Completion 2027-05-02 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety level on the Beck Anxiety Inventory (BAI) from baseline to 12 months after therapy | T1: Baseline (before the intervention); T2: 5 weeks (mid-intervention); T3: 10 weeks (immediately after the intervention); T4: 22 weeks (3 months after the intervention); T5: 34 weeks (6 months after the intervention); T6: 60 weeks (12 months after)
  Total score on the Beck Anxiety Inventory (BAI). The scale consists of 21 items, where each item is rated from 0 to 3 points. The total score ranges from 0 to 63. A higher score indicates a higher level of anxiety (0-7: minimal, 8-15: mild, 16-25: moderate, 26-63: severe anxiety)
Change in Hospital Anxiety and Depression Scale - Anxiety (HADS-A) subscale scores from baseline to 12 months after therapy | T1: Baseline (before the intervention); T2: 5 weeks (mid-intervention); T3: 10 weeks (immediately after the intervention); T4: 22 weeks (3 months after the intervention); T5: 34 weeks (6 months after the intervention); T6: 60 weeks (12 months after)
  Total score for the HADS-A anxiety subscale. The subscale contains 7 questions, each of which is scored from 0 to 3 points. The total score ranges from 0 to 21. A higher score indicates a higher level of anxiety (0-7: normal, 8-10: subclinically expressed anxiety, 11-21: clinically expressed anxiety)
Change in total score according to the "I - Reconstruction" diagnosis of preverbal dysregulation (DPD) method from baseline to 12 months after therapy | T1: Baseline (before the intervention); T2: 5 weeks (mid-intervention); T3: 10 weeks (immediately after the intervention); T4: 22 weeks (3 months after the intervention); T5: 34 weeks (6 months after the intervention); T6: 60 weeks (12 months after)
  A general measure of the level of preverbal trauma, including three scales: possession, pleasure, and desire. Each scale contains 3 questions. The total score ranges from 0 to 45. A higher score indicates a higher degree of severity of preverbal trauma

SECONDARY OUTCOMES:
Change in depression scores on the Beck Depression Inventory (BDI) from baseline to 12 months after intervention | T1: Baseline (before the intervention); T2: 5 weeks (mid-intervention); T3: 10 weeks (immediately after the intervention); T4: 22 weeks (3 months after the intervention); T5: 34 weeks (6 months after the intervention); T6: 60 weeks (12 months after)
  Total score on the BDI-II questionnaire, consisting of 21 items. Each response is scored from 0 to 3 points. The total score ranges from 0 to 63. Higher scores indicate higher severity of depressive symptoms (0-13: minimal, 14-19: mild, 20-28: moderate, 29-63: severe depression)
Change in Hospital Anxiety and Depression Scale (HADS-D) Depression subscale scores from baseline to 12 months post-intervention | T1: Baseline (before the intervention); T2: 5 weeks (mid-intervention); T3: 10 weeks (immediately after the intervention); T4: 22 weeks (3 months after the intervention); T5: 34 weeks (6 months after the intervention); T6: 60 weeks (12 months after)
  Total score on the HADS-D depression subscale (7 questions). Each response is scored from 0 to 3 points. The total score ranges from 0 to 21. A higher score indicates a higher level of depressive symptoms (0-7: normal, 8-10: subclinical depression, 11-21: clinical depression)
Change in the level of internal conflicts according to the "Internal Conflict Test" from baseline to 12 months after intervention | T1: Baseline (before the intervention); T2: 5 weeks (mid-intervention); T3: 10 weeks (immediately after the intervention); T4: 22 weeks (3 months after the intervention); T5: 34 weeks (6 months after the intervention); T6: 60 weeks (12 months after)
  In the "Internal Conflict Test" questionnaire, the indicator is measured in points. From 0 to 27. A higher score indicates a higher level of intensity of internal conflicts.

CONTACTS AND LOCATIONS:
Overall Officials: Tetiana Pavlenko, Principal Investigator — International Association of Psychosomatics and Health Therapy
Locations (1):
- International Association of Psychosomatics and Body Therapy, Kyiv, Kyiv Oblast, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
Depersonalized individual participant data (IPD) will be shared, including demographic characteristics (e.g., age, gender), results of psychometric assessments collected at specified time points in the study, and information on participant assignment to study groups and adherence to the intervention protocol. The data will not contain any direct or indirect personal identifiers. The amount of IPD shared will be limited to variables necessary to reproduce the primary and secondary analyses published in scientific journals and will comply with data minimization principles and ethical and regulatory oversight requirements.
Supporting Information: Study Protocol, SAP, ICF
Access Criteria: Access to individual depersonalized participant data (IPD) and related supporting information may be provided to independent researchers after publication of the main results of the study in specialized scientific journals. Access will be granted exclusively on the basis of a substantiated scientific request, containing a clearly defined purpose of data use, an analysis plan and confirmation of compliance with ethical principles. The volume of accessible data will be limited to depersonalized sets of IPD and relevant methodological documentation (e.g. description of variables and study protocol). Data transfer will be carried out in accordance with applicable data exchange agreements and subject to full compliance with ethical and regulatory requirements that guarantee the confidentiality and protection of personal information of participants.

REFERENCES:
- See also: Lifetime prevalence and distribution of mental disorders by age of onset in the World Health Organization's Global Mental Health Survey Initiative — https://pubmed.ncbi.nlm.nih.gov/18188442/
- See also: The global burden of mental disorders: updated data from the WHO World Mental Health Survey (WMH) — https://pubmed.ncbi.nlm.nih.gov/19378696/
- See also: World Federation of Societies of Biological Psychiatry (WFSBP) guidelines for treatment of anxiety, obsessive-compulsive and posttraumatic stress disorders - Version 3. Part I: Anxiety disorders — https://pubmed.ncbi.nlm.nih.gov/35900161/
- See also: How Much Does Therapy Cost in Zurich? 2025 Guide — https://www.therapyroute.com/article/how-much-does-therapy-cost-in-zurich-2025-guide-by-therapyroute
- See also: Kernberg, O. F. (1993). The current status of psychoanalysis. Journal of the American Psychoanalytic Association, 41(1), 45-62. — https://www.therapyroute.com/article/how-much-does-therapy-cost-in-zurich-2025-guide-by-therapyroute
- See also: Retrospective Analysis of Mental Disorder Patients with "Combination of Medical Care and Nursing Care" — https://www.scirp.org/reference/referencespapers?referenceid=3268701
- See also: The Mental Health Implications of a Local Epidemic: Early Experience with the COVID-19 Outbreak in Wuhan — https://www.scirp.org/reference/referencespapers?referenceid=2907885
- See also: Anhedonia and anxiety underlying depressive symptomatology have distinct effects on reward-based decision-making — https://doi.org/10.1371/journal.pone.0186473
- See also: Reconsidering anhedonia in depression: Lessons from translational neuroscience — https://www.researchgate.net/publication/45094186_Treadway_MT_Zald_DH_Reconsidering_anhedonia_in_depression_Lessons_from_translational_neuroscience_Neurosci_Biobehav_Rev_35_537-555